CLINICAL TRIAL: NCT01378377
Title: Phase I Dose Escalation Trial of MEK1/2 Inhibitor MSC1936369B Combined With Temsirolimus in Subjects With Advanced Solid Tumors
Brief Title: Combination Trial of Pimasertib (MSC1936369B) With Temsirolimus
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was stopped due to the toxicities observed with the combination of pimasertib and temsirolimus.
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 200066-005
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2017-10

CONDITIONS: Advanced Solid Tumor
Keywords: MEK inhibitor; Temsirolimus; Neoplasms; Phase I; Pimasertib
MeSH Terms: conditions — Neoplasms | interventions — N-(2,3-dihydroxypropyl)-1-((2-fluoro-4-iodophenyl)amino)isonicotinamide; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pimasertib 45 mg+Temsirolimus 12.5 mg (Experimental)
  Interventions: Drug: Pimasertib; Drug: Temsirolimus
- Pimasertib 45 mg+Temsirolimus 25 mg (Experimental)
  Interventions: Drug: Pimasertib; Drug: Temsirolimus
- Pimasertib 75 mg+Temsirolimus 25 mg (Experimental)
  Interventions: Drug: Pimasertib; Drug: Temsirolimus

INTERVENTIONS:
Drug: Pimasertib — Pimasertib will be administered in fasted state at a dose of 45 mg once daily orally on Days 1 to 15. Treatment will be continued until disease progression, intolerable toxicity, investigator's decision to discontinue treatment, or withdrawal of consent.
  Other Names: MSC1936369B
  Arms: Pimasertib 45 mg+Temsirolimus 12.5 mg; Pimasertib 45 mg+Temsirolimus 25 mg
Drug: Pimasertib — Pimasertib will be administered in fasted state at a dose of 75 mg once daily orally on Days 1 to 15. Treatment will be continued until disease progression, intolerable toxicity, investigator's decision to discontinue treatment, or withdrawal of consent.
  Other Names: MSC1936369B
  Arms: Pimasertib 75 mg+Temsirolimus 25 mg
Drug: Temsirolimus — Temsirolimus will be administered at a dose of 12.5 mg as intravenous infusion over a 30-60 minute period once a week within 10 minutes after administration of pimasertib on Days 1, 8 and 15 in successive 21-day cycles. Treatment will be continued until disease progression, intolerable toxicity, investigator's decision to discontinue treatment, or withdrawal of consent.
  Arms: Pimasertib 45 mg+Temsirolimus 12.5 mg
Drug: Temsirolimus — Temsirolimus will be administered at a dose of 25 mg as intravenous infusion over a 30-60 minute period once a week within 10 minutes after administration of pimasertib on Days 1, 8 and 15 in successive 21-day cycles. Treatment will be continued until disease progression, intolerable toxicity, investigator's decision to discontinue treatment, or withdrawal of consent.
  Arms: Pimasertib 45 mg+Temsirolimus 25 mg; Pimasertib 75 mg+Temsirolimus 25 mg

SUMMARY:
The research trial is testing the experimental drug pimasertib and the drug Torisel, given together, in the treatment of advanced solid tumors. The primary purpose of the study is to determine the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D) of the drug combination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically or cytologically confirmed solid tumors, either refractory to standard therapy or for which no effective standard therapy is available.
* Measurable or evaluable disease at baseline by RECIST 1.0.
* Age >= 18 years.
* Subject has read and understands the informed consent form and is willing and able to give informed consent.
* Performance Status score of less than or equal to (<=) 1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
* Women of childbearing potential must have a negative blood pregnancy test at the screening visit.
* Female subjects of childbearing potential and male subjects with female partners of childbearing potential must be willing to avoid pregnancy by using an adequate method of contraception for 2 weeks prior to screening, during the trial and for 3 months after the last dose of trial medication.

Additional inclusion criteria also apply.

Exclusion Criteria:

* The subject has previously been treated with mammalian target of rapamycin (mTOR) inhibitor or a mitogen-activated protein kinase (MEK) inhibitor and taken off treatment due to drug-related AEs.
* The subject has received any of the following:
* Chemotherapy, immunotherapy, hormonal therapy, biologic therapy, any investigational agent or any other anti-cancer therapy within 28 days (6 weeks for nitrosoureas or mitomycin C) of Day 1 of trial treatment; non-cytotoxic chemotherapy or investigational agent with limited potential for delayed toxicity is permitted if terminated at least 5 half-lives prior to Day 1 of trial treatment.
* Extensive prior radiotherapy on more than 30% of bone marrow reserves, or prior bone marrow/stem cell transplantation.
* The subject has not recovered from toxicity due to prior therapy to baseline or CTCAE v4.0 of Grade 1 or less (except alopecia).
* The subject has poor organ or marrow function as defined in protocol.
* History of central nervous system (CNS) metastases or primary CNS tumor, unless subject has been previously treated for these conditions, is asymptomatic and has had no requirement for anticonvulsants or high dose corticosteroids for a minimum of 2 weeks prior to entry into the trial.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months of Day 1 of trial drug treatment.
* Recent major surgery or trauma (within the last 28 days), unhealing/open wounds, diabetic ulcers, recent drainage of significant volume of ascites or pleural effusion.
* History of congestive heart failure, unstable angina, myocardial infarction, symptomatic cardiac conduction abnormality, pacemaker, or other clinically significant cardiac disease or history of a stroke within 3 months prior to entering the trial.
* Baseline corrected QT interval on screening electrocardiogram (ECG) (QTc) >= 460 ms or left ventricular ejection fraction (LVEF) < 40% on screening echocardiogram.
* Other uncontrolled intercurrent diseases
* Retinal degenerative disease (hereditary retinal degeneration or age-related macular degeneration), history of uveitis or history of retinal vein occlusion, or medically relevant abnormal ophthalmology assessments at screening.
* Known or suspected allergy to pimasertib, temsirolimus, other rapamycins (sirolimus, everolimus, etc.), their excipients, or any agent given in the course of this trial.
* Immunization with attenuated live vaccines within one week of trial entry (examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, etc.).
* Concomitant use of any medications or substances that are strong inhibitors or inducers of CYP3A enzyme, including, but not limited to, phenytoin, carbamazepine, barbiturates, azoles, rifampin, phenobarbital, or St. John's Wort.
* Pregnant or lactating female.
* Legal incapacity or limited legal capacity.

Additional exclusion criteria also apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-05-27 (Actual); Primary Completion 2012-02-23 (Actual); Study Completion 2012-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono, an affiliate of MerckKGaA, Darmstadt, Germany
Locations (3):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - For Recruiting Locations in the US contact US Medical Information in, Rockland, Massachusetts
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Mita M, Fu S, Piha-Paul SA, Janku F, Mita A, Natale R, Guo W, Zhao C, Kurzrock R, Naing A. Phase I trial of MEK 1/2 inhibitor pimasertib combined with mTOR inhibitor temsirolimus in patients with advanced solid tumors. Invest New Drugs. 2017 Oct;35(5):616-626. doi: 10.1007/s10637-017-0442-3. Epub 2017 Feb 13. PMID 28194539
- [Derived] Liu X, Lorusso P, Mita M, Piha-Paul S, Hong DS, Fu S, McQuinn L, Asatiani E, Doyle LA, Chen HX, Hess KR, Kurzrock R, Naing A. Incidence of mucositis in patients treated with temsirolimus-based regimens and correlation to treatment response. Oncologist. 2014 Apr;19(4):426-8. doi: 10.1634/theoncologist.2013-0231. Epub 2014 Mar 25. PMID 24668327

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last subject (informed consent): 27 May 2011/23 August 2012. Last subject completed: 23 February 2012; Subjects randomized at 2 centers in United States.
Pre-assignment Details: 46 screened for eligibility; 13 were excluded (mainly non-fulfillment of inclusion or exclusion criteria). 33 subjects were enrolled and treated in the study.
Groups:
- Pimasertib 45 mg+Temsirolimus 12.5 mg: Pimasertib was administered in fasted state at a dose of 45 mg once daily orally on Days 1 to 15. Temsirolimus was administered at a dose of 12.5 mg as intravenous infusion over a 30-60 minute period once a week within 10 minutes after administration of pimasertib on Days 1, 8 and 15 in successive 21-day cycles. Treatment was continued until disease progression, intolerable toxicity, investigator's decision to discontinue treatment, or withdrawal of consent.
- Pimasertib 45 mg+Temsirolimus 25 mg: Pimasertib was administered in fasted state at a dose of 45 mg once daily orally on Days 1 to 15. Temsirolimus was administered at a dose of 25 mg as intravenous infusion over a 30-60 minute period once a week within 10 minutes after administration of pimasertib on Days 1, 8 and 15 in successive 21-day cycles. Treatment was continued until disease progression, intolerable toxicity, investigator's decision to discontinue treatment, or withdrawal of consent.
- Pimasertib 75 mg+Temsirolimus 25 mg: Pimasertib was administered in fasted state at a dose of 75 mg once daily orally on Days 1 to 15. Temsirolimus was administered at a dose of 25 mg as intravenous infusion over a 30-60 minute period once a week within 10 minutes after administration of pimasertib on Days 1, 8 and 15 in successive 21-day cycles. Treatment was continued until disease progression, intolerable toxicity, investigator's decision to discontinue treatment, or withdrawal of consent.
Period: Overall Study
Arm/Group | Pimasertib 45 mg+Temsirolimus 12.5 mg | Pimasertib 45 mg+Temsirolimus 25 mg | Pimasertib 75 mg+Temsirolimus 25 mg
Started | 4 | 23 | 6
Completed | 4 | 23 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all the subjects who received at least one administration of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pimasertib 45 mg+Temsirolimus 12.5 mg | Pimasertib 45 mg+Temsirolimus 25 mg | Pimasertib 75 mg+Temsirolimus 25 mg | Total
Number analyzed (Participants) | 4 | 23 | 6 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (11.30) | 57.9 (14.09) | 55.5 (6.19) | 58.1 (12.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 16 | 4 | 22
  Male | 2 | 7 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Dose Limiting Toxicities (DLTs)
Description: DLT was defined as any of the following toxicities graded as per National Cancer Institute (NCI) common terminology criteria for adverse events (NCI CTCAE v4.0) encountered within cycle 1 of treatment at any dose level and judged not to be related to the underlying disease or concomitant medications. A treatment emergent adverse event (TEAE) of potential clinical significance such that further dose escalation would expose subjects to unacceptable risk; any Grade >=3 non-hematological toxicity except Grade 3 asymptomatic increases in liver function tests, diarrhea, nausea or vomiting with duration <= 48 hours and alopecia; Grade 4 neutropenia of >5 days duration or febrile neutropenia of >1 day duration; Grade 3 thrombocytopenia with bleeding or Grade 4 thrombocytopenia; any treatment interruption >2 weeks due to adverse events; any severe, impairing daily functions or life-threatening, complication or abnormality not defined in NCI-CTCAE that is attributable to the therapy.
Time Frame: Up to 21 Days (within Cycle 1)
Population: The dose escalation analysis set included all the subjects who received at least 80% of the planned doses of each treatment (pimasertib and temsirolimus) in the first cycle of treatment or who experienced DLT during the first cycle of treatment regardless of the received amount of drug.
Measure: Number; unit: subjects
Arm/Group | Pimasertib 45 mg+Temsirolimus 12.5 mg | Pimasertib 45 mg+Temsirolimus 25 mg | Pimasertib 75 mg+Temsirolimus 25 mg
Number analyzed (Participants) | 3 | 17 | 6
subjects | 0 | 7 | 2

2. Secondary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs)
Description: An AE was defined as any new untoward medical occurrences/worsening of pre-existing medical condition, whether or not related to study drug. The TEAEs were those events that occur between first dose of trial treatment and up to 30 days after last dose of the trial treatment that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From the start of the trial treatment until data cut-off date (23 February 2012)
Population: The safety analysis set included all the subjects who received at least one administration of trial medication.
Measure: Number; unit: subjects
Arm/Group | Pimasertib 45 mg+Temsirolimus 12.5 mg | Pimasertib 45 mg+Temsirolimus 25 mg | Pimasertib 75 mg+Temsirolimus 25 mg
Number analyzed (Participants) | 4 | 23 | 6
subjects | 4 | 23 | 6

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Pimasertib
Description: Pharmacokinetic parameters were reported based on DDI and non-DDI cohorts as per plan.
Time Frame: Drug-drug interaction (DDI) cohorts: Days 1 and 9 of Cycle 1; Non-DDI cohorts: Day 8 of Cycle 1
Population: Pharmacokinetic analysis was performed in all the subjects who received at least one administration of trial medication and whose plasma samples were collected. "Number Analyzed" signifies subjects evaluable for this measure for specified categories for each reporting group, respectively.
Measure: Median (Full Range); unit: nanogram/milliliter
Groups:
- Pimasertib 45 mg+Temsirolimus 12.5 mg (DDI): Pimasertib was administered in fasted state at a dose of 45 mg once daily orally on Days 1 to 15. Temsirolimus was administered at a dose of 12.5 mg as intravenous infusion over a 30-60 minute period once a week within 10 minutes after administration of pimasertib on Days 1, 8 and 15 in successive 21-day cycles. Treatment was continued until disease progression, intolerable toxicity, investigator's decision to discontinue treatment, or withdrawal of consent. Subjects were analyzed for drug-drug interaction.
- Pimasertib 45 mg+Temsirolimus 25 mg (DDI): Pimasertib was administered in fasted state at a dose of 45 mg once daily orally on Days 1 to 15. Temsirolimus was administered at a dose of 25 mg as intravenous infusion over a 30-60 minute period once a week within 10 minutes after administration of pimasertib on Days 1, 8 and 15 in successive 21-day cycles. Treatment was continued until disease progression, intolerable toxicity, investigator's decision to discontinue treatment, or withdrawal of consent. Subjects were analyzed for drug-drug interaction.
- Pimasertib 45 mg+Temsirolimus 25 mg (Non-DDI): Pimasertib was administered in fasted state at a dose of 45 mg once daily orally on Days 1 to 15. Temsirolimus was administered at a dose of 25 mg as intravenous infusion over a 30-60 minute period once a week within 10 minutes after administration of pimasertib on Days 1, 8 and 15 in successive 21-day cycles. Treatment was continued until disease progression, intolerable toxicity, investigator's decision to discontinue treatment, or withdrawal of consent. Subjects were not analyzed for drug-drug interaction.
- Pimasertib 75 mg+Temsirolimus 25 mg (Non-DDI): Pimasertib was administered in fasted state at a dose of 75 mg once daily orally on Days 1 to 15. Temsirolimus was administered at a dose of 25 mg as intravenous infusion over a 30-60 minute period once a week within 10 minutes after administration of pimasertib on Days 1, 8 and 15 in successive 21-day cycles. Treatment was continued until disease progression, intolerable toxicity, investigator's decision to discontinue treatment, or withdrawal of consent. Subjects were not analyzed for drug-drug interaction.
Arm/Group | Pimasertib 45 mg+Temsirolimus 12.5 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (Non-DDI) | Pimasertib 75 mg+Temsirolimus 25 mg (Non-DDI)
Number analyzed (Participants) | 4 | 15 | 5 | 6
nanogram/milliliter
  DDI: Day 1: number analyzed (Participants) | 4 | 15 | 0 | 0
  DDI: Day 1 | 185.2 [87.38 to 266.5] | 193.5 [97.24 to 326.5] |  |
  DDI: Day 9: number analyzed (Participants) | 4 | 13 | 0 | 0
  DDI: Day 9 | 131 [68.75 to 190.5] | 192.1 [63.8 to 406] |  |
  Non-DDI: Day 8: number analyzed (Participants) | 0 | 0 | 5 | 6
  Non-DDI: Day 8 |  |  | 197.6 [73.75 to 317.3] | 308.1 [157.3 to 460]

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Temsirolimus
Description: Pharmacokinetic parameters were reported based on DDI and non-DDI cohorts as per plan.
Time Frame: DDI cohorts: Days 9 and 16 of Cycle 1; Non-DDI cohorts: Day 8 of Cycle 8
Population: as for outcome 3
Measure: Median (Full Range); unit: nanogram/milliliter
Arm/Group | Pimasertib 45 mg+Temsirolimus 12.5 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (Non-DDI) | Pimasertib 75 mg+Temsirolimus 25 mg (Non-DDI)
Number analyzed (Participants) | 4 | 10 | 4 | 6
nanogram/milliliter
  DDI: Day 9: number analyzed (Participants) | 4 | 10 | 0 | 0
  DDI: Day 9 | 457.5 [361.6 to 578.1] | 505.3 [396.8 to 591.4] |  |
  DDI: Day 16: number analyzed (Participants) | 3 | 4 | 0 | 0
  DDI: Day 16 | 281.1 [13.21 to 636.4] | 511.8 [184.6 to 575.9] |  |
  Non-DDI: Day 8: number analyzed (Participants) | 0 | 0 | 4 | 6
  Non-DDI: Day 8 |  |  | 489.9 [391.9 to 525.5] | 480.9 [323.3 to 589.7]

5. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Pimasertib
Description: Pharmacokinetic parameters were reported based on DDI and non-DDI cohorts as per plan.
Time Frame: DDI cohorts: Days 1 and 9 of Cycle 1; Non-DDI cohorts: Day 8 of Cycle 1
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Pimasertib 45 mg+Temsirolimus 12.5 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (Non-DDI) | Pimasertib 75 mg+Temsirolimus 25 mg (Non-DDI)
Number analyzed (Participants) | 4 | 15 | 5 | 6
hour
  DDI: Day 1: number analyzed (Participants) | 4 | 15 | 0 | 0
  DDI: Day 1 | 1 [0.5333 to 2] | 1.5 [0 to 4] |  |
  DDI: Day 9: number analyzed (Participants) | 4 | 13 | 0 | 0
  DDI: Day 9 | 2.3 [0.9167 to 4.033] | 1.133 [0.5 to 2.667] |  |
  Non-DDI: Day 8: number analyzed (Participants) | 0 | 0 | 5 | 6
  Non-DDI: Day 8 |  |  | 1.5 [1 to 3.967] | 0.5833 [0.5 to 3]

6. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Temsirolimus
Description: Pharmacokinetic parameters were reported based on DDI and non-DDI cohorts as per plan.
Time Frame: DDI cohorts: Days 9 and 16 of Cycle 1; Non-DDI cohorts: Day 8 of Cycle 1
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Pimasertib 45 mg+Temsirolimus 12.5 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (Non-DDI) | Pimasertib 75 mg+Temsirolimus 25 mg (Non-DDI)
Number analyzed (Participants) | 4 | 10 | 4 | 6
hour
  DDI: Day 9: number analyzed (Participants) | 4 | 10 | 0 | 0
  DDI: Day 9 | 0.7417 [0.5167 to 1] | 0.5667 [0.5 to 1.017] |  |
  DDI: Day 16: number analyzed (Participants) | 3 | 4 | 0 | 0
  DDI: Day 16 | 0.9333 [0.5 to 24.05] | 0.5 [0.5 to 1.55] |  |
  Non-DDI: Day 8: number analyzed (Participants) | 0 | 0 | 4 | 6
  Non-DDI: Day 8 |  |  | 0.5 [0.5 to 0.55] | 0.55 [0.4333 to 0.5833]

7. Secondary Outcome: Area Under the Concentration Time Curve During a Dosing Interval (AUCtau) and Area Under the Concentration Time Curve From Time Zero to Infinity (AUC0-inf) of Pimasertib
Description: The AUCtau was defined as the area under the concentration curve divided by the dosing interval. AUC(0-inf) was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity. Pharmacokinetic parameters were reported based on DDI and non-DDI cohorts as per plan.
Time Frame: DDI cohorts: Days 9 of Cycle 1; Non-DDI cohorts: Day 8 of Cycle 1 for AUCtau; DDI cohorts: Day 1 of Cycle 1 AUC0-inf
Population: Pharmacokinetic analysis was performed in all the subjects who received at least one administration of trial medication and whose plasma samples were collected. 'N'=subjects evaluable for this outcome measure; "Number Analyzed" signifies subjects evaluable for this measure for specified categories for each reporting group, respectively.
Measure: Median (Full Range); unit: hour*nanogram/milliliter
Arm/Group | Pimasertib 45 mg+Temsirolimus 12.5 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (Non-DDI) | Pimasertib 75 mg+Temsirolimus 25 mg (Non-DDI)
Number analyzed (Participants) | 4 | 14 | 4 | 6
hour*nanogram/milliliter
  DDI: AUCtau: Day 9: number analyzed (Participants) | 4 | 13 | 0 | 0
  DDI: AUCtau: Day 9 | 628 [435.6 to 1338] | 805 [264.3 to 1623] |  |
  Non-DDI: AUCtau: Day 8: number analyzed (Participants) | 0 | 0 | 4 | 6
  Non-DDI: AUCtau: Day 8 |  |  | 706 [333.8 to 2548] | 1402 [922.2 to 1735]
  DDI: AUC0-inf: Day 1: number analyzed (Participants) | 4 | 14 | 0 | 0
  DDI: AUC0-inf: Day 1 | 573.2 [393.5 to 1703] | 828.6 [373.3 to 1310] |  |

8. Secondary Outcome: Area Under Plasma Concentration Time Curve From Time Zero to Infinity (AUC0-inf) of Temsirolimus
Description: The AUC(0-inf) was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity. Pharmacokinetic parameters were reported based on DDI and non-DDI cohorts as per plan.
Time Frame: DDI cohorts: Days 9 and 16 of Cycle 1; Non-DDI cohorts: Day 8 of Cycle 1
Population: Pharmacokinetic analysis was performed in all the subjects who received at least one administration of trial medication and whose plasma samples were collected. 'N'=subjects evaluable for this outcome measure;"Number Analyzed" signifies subjects evaluable for this measure for specified categories for each reporting group, respectively.
Measure: Median (Full Range); unit: hour*nanogram/milliliter
Arm/Group | Pimasertib 45 mg+Temsirolimus 12.5 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (Non-DDI) | Pimasertib 75 mg+Temsirolimus 25 mg (Non-DDI)
Number analyzed (Participants) | 4 | 10 | 4 | 5
hour*nanogram/milliliter
  DDI: Day 9: number analyzed (Participants) | 4 | 10 | 0 | 0
  DDI: Day 9 | 2452 [1670 to 4440] | 2130 [1534 to 3642] |  |
  DDI: Day 16: number analyzed (Participants) | 2 | 4 | 0 | 0
  DDI: Day 16 | 2006 [1174 to 2837] | 2743 [1977 to 3219] |  |
  Non-DDI: Day 8: number analyzed (Participants) | 0 | 0 | 4 | 5
  Non-DDI: Day 8 |  |  | 4026 [2386 to 4783] | 2194 [1324 to 2483]

9. Secondary Outcome: Apparent Terminal Half-life (t1/2) of Pimasertib
Description: The t1/2 was defined as the time required for the plasma concentration of drug to decrease 50% in the final stage of its elimination. Pharmacokinetic parameters were reported based on DDI and non-DDI cohorts as per plan.
Time Frame: DDI cohorts: Days 1 and 9 of Cycle 1; Non-DDI cohorts: Day 8 of Cycle 1
Population: as for outcome 7
Measure: Median (Full Range); unit: hour
Arm/Group | Pimasertib 45 mg+Temsirolimus 12.5 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (Non-DDI) | Pimasertib 75 mg+Temsirolimus 25 mg (Non-DDI)
Number analyzed (Participants) | 4 | 14 | 4 | 6
hour
  DDI: Day 1: number analyzed (Participants) | 4 | 14 | 0 | 0
  DDI: Day 1 | 5.915 [4.718 to 6.652] | 5.886 [2.504 to 20.25] |  |
  DDI: Day 9: number analyzed (Participants) | 4 | 13 | 0 | 0
  DDI: Day 9 | 6.08 [2.101 to 11.17] | 5.896 [2.013 to 23.86] |  |
  Non-DDI: Day 8: number analyzed (Participants) | 0 | 0 | 4 | 6
  Non-DDI: Day 8 |  |  | 7.746 [5.625 to 9.993] | 5.712 [2.365 to 8.656]

10. Secondary Outcome: Apparent Terminal Half-life (t1/2) of Temsirolimus
Description: as for outcome 9
Time Frame: DDI cohorts: Days 9 and 16 of Cycle 1; Non-DDI cohorts: Day 8 of Cycle 1
Population: Pharmacokinetic analysis was performed in all the subjects who received at least one administration of trial medication and whose plasma samples were collected. N=subjects evaluable for this outcome measure; "Number Analyzed" signifies subjects evaluable for this measure for specified categories for each reporting group, respectively.
Measure: Median (Full Range); unit: hour
Arm/Group | Pimasertib 45 mg+Temsirolimus 12.5 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (Non-DDI) | Pimasertib 75 mg+Temsirolimus 25 mg (Non-DDI)
Number analyzed (Participants) | 4 | 10 | 4 | 5
hour
  DDI: Day 9: number analyzed (Participants) | 4 | 10 | 0 | 0
  DDI: Day 9 | 25.57 [10.39 to 54.46] | 13.2 [9.237 to 34.92] |  |
  DDI: Day 16: number analyzed (Participants) | 2 | 4 | 0 | 0
  DDI: Day 16 | 20.62 [12.97 to 28.27] | 19.14 [13.54 to 25.82] |  |
  Non-DDI: Day 8: number analyzed (Participants) | 0 | 0 | 4 | 5
  Non-DDI: Day 8 |  |  | 29.08 [26.14 to 44.14] | 10.42 [9.192 to 13.76]

11. Secondary Outcome: Apparent Clearance From Plasma Following Oral Administration (CL/f) of Pimasertib
Description: Clearance (CL) of a drug was a measure of the rate at which a drug was metabolized or eliminated by normal biological processes. The CL obtained after oral dose (CL/F) was influenced by the fraction of the dose absorbed (bioavailability). Pharmacokinetic parameters were reported based on DDI and non-DDI cohorts as per plan.
Time Frame: DDI cohorts: Days 1 and 9 of Cycle 1; Non-DDI cohorts: Day 8 of Cycle 1
Population: Pharmacokinetic analysis was performed in all the subjects who received at least one administration of trial medication and whose plasma samples were collected. 'N' =subjects evaluable for this outcome measure;"Number Analyzed" signifies subjects evaluable for this measure for specified categories for each reporting group, respectively.
Measure: Median (Full Range); unit: liter/hour
Arm/Group | Pimasertib 45 mg+Temsirolimus 12.5 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (Non-DDI) | Pimasertib 75 mg+Temsirolimus 25 mg (Non-DDI)
Number analyzed (Participants) | 4 | 14 | 4 | 6
liter/hour
  DDI: Day 1: number analyzed (Participants) | 4 | 14 | 0 | 0
  DDI: Day 1 | 81.25 [26.42 to 114.4] | 54.36 [34.36 to 120.6] |  |
  DDI: Day 9: number analyzed (Participants) | 4 | 13 | 0 | 0
  DDI: Day 9 | 71.99 [33.63 to 103.3] | 55.9 [27.73 to 170.3] |  |
  Non-DDI: Day 8: number analyzed (Participants) | 0 | 0 | 4 | 6
  Non-DDI: Day 8 |  |  | 64.31 [17.66 to 134.8] | 53.6 [43.22 to 81.33]

12. Secondary Outcome: Total Body Clearance From Plasma Following Intravenous Administration (CL) of Temsirolimus
Description: The clearance of a drug was a measure of the rate at which a drug was metabolized or eliminated by normal biological processes. Pharmacokinetic parameters were reported based on DDI and non-DDI cohorts as per plan.
Time Frame: DDI cohorts: Days 9 and 16 of Cycle 1; Non-DDI cohorts: Day 8 of Cycle 1
Population: Pharmacokinetic analysis was performed in all the subjects who received at least one administration of trial medication and whose plasma samples were collected. 'N' =subjects evaluable for this outcome measure; "Number Analyzed" signifies subjects evaluable for this measure for specified categories for each reporting group, respectively.
Measure: Median (Full Range); unit: liter/hour
Arm/Group | Pimasertib 45 mg+Temsirolimus 12.5 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (Non-DDI) | Pimasertib 75 mg+Temsirolimus 25 mg (Non-DDI)
Number analyzed (Participants) | 4 | 10 | 4 | 5
liter/hour
  DDI: Day 9: number analyzed (Participants) | 4 | 10 | 0 | 0
  DDI: Day 9 | 5.378 [2.815 to 7.486] | 11.73 [6.863 to 16.29] |  |
  DDI: Day 16: number analyzed (Participants) | 2 | 4 | 0 | 0
  DDI: Day 16 | 7.528 [4.406 to 10.65] | 9.292 [7.766 to 12.64] |  |
  Non-DDI: Day 8: number analyzed (Participants) | 0 | 0 | 4 | 5
  Non-DDI: Day 8 |  |  | 6.284 [5.227 to 10.48] | 11.39 [10.07 to 18.89]

13. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Pimasertib
Description: Volume of distribution (Vz) was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. The Vz after oral dose (Vz/F) was influenced by the fraction absorbed. Pharmacokinetic parameters were reported based on DDI and non-DDI cohorts as per plan.
Time Frame: DDI cohorts: Days 1 and 9 of Cycle 1; Non-DDI cohorts: Day 8 of Cycle 1
Population: as for outcome 12
Measure: Median (Full Range); unit: liter
Groups:
- Pimasertib 75 mg+Temsirolimus (TEM) 25 mg (Non-DDI): Pimasertib was administered in fasted state at a dose of 75 mg once daily orally on Days 1 to 15. Temsirolimus was administered at a dose of 25 mg as intravenous infusion over a 30-60 minute period once a week within 10 minutes after administration of pimasertib on Days 1, 8 and 15 in successive 21-day cycles. Treatment was continued until disease progression, intolerable toxicity, investigator's decision to discontinue treatment, or withdrawal of consent. Subjects were not analyzed for drug-drug interaction.
Arm/Group | Pimasertib 45 mg+Temsirolimus 12.5 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (Non-DDI) | Pimasertib 75 mg+Temsirolimus (TEM) 25 mg (Non-DDI)
Number analyzed (Participants) | 4 | 14 | 4 | 6
liter
  DDI: Day 1: number analyzed (Participants) | 4 | 14 | 0 | 0
  DDI: Day 1 | 691.3 [210.3 to 923] | 536.5 [199.4 to 1450] |  |
  DDI: Day 9: number analyzed (Participants) | 4 | 13 | 0 | 0
  DDI: Day 9 | 517.6 [274.4 to 1080] | 519.5 [157.3 to 1768] |  |
  Non-DDI: Day 8: number analyzed (Participants) | 0 | 0 | 4 | 6
  Non-DDI: Day 8 |  |  | 760.6 [143.3 to 1840] | 416.5 [190.4 to 745.5]

14. Secondary Outcome: Volume of Distribution (Vz) of Temsirolimus
Description: The Vz was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Pharmacokinetic parameters were reported based on DDI and non-DDI cohorts as per plan.
Time Frame: DDI cohorts: Days 9 and 16 of Cycle 1; Non-DDI cohorts: Day 8 of Cycle 1
Population: as for outcome 3
Measure: Median (Full Range); unit: liter
Arm/Group | Pimasertib 45 mg+Temsirolimus 12.5 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (Non-DDI) | Pimasertib 75 mg+Temsirolimus 25 mg (Non-DDI)
Number analyzed (Participants) | 4 | 10 | 4 | 5
liter
  DDI: Day 9: number analyzed (Participants) | 4 | 10 | 0 | 0
  DDI: Day 9 | 152 [99.01 to 326.1] | 244.5 [142.2 to 505.4] |  |
  DDI: Day 16: number analyzed (Participants) | 2 | 4 | 0 | 0
  DDI: Day 16 | 189.5 [179.6 to 199.3] | 233 [216.1 to 394.4] |  |
  Non-DDI: Day 8: number analyzed (Participants) | 0 | 0 | 4 | 5
  Non-DDI: Day 8 |  |  | 309.7 [203.6 to 471.3] | 172.9 [133.5 to 375]

15. Secondary Outcome: Number of Subjects With Disease Control Rate
Description: Disease control is defined as confirmed complete response (CR), partial response (PR), or stable disease (SD) >=12 weeks), based on tumor assessments as determined by Response Evaluation Criteria In Solid Tumors (RECIST) version 1.0. CR: The disappearance of all lesions and normalization of tumor marker level. PR: At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the sum of the longest diameter at baseline. SD: Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum of the longest diameter since treatment started.
Time Frame: From the start of the trial treatment until data cut-off date (23 February 2012)
Population: Data was not evaluated for this outcome as the subjects did not met the minimum criteria duration for the evaluation of the outcome measure due to the early termination of the trial
Arm/Group | Pimasertib 45 mg+Temsirolimus 12.5 mg | Pimasertib 45 mg+Temsirolimus 25 mg | Pimasertib 75 mg+Temsirolimus 25 mg
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Phospho Extracellular Signal Regulated Kinase (pERK ) Levels and Phospho Ribosomal Protein S6 (pS6) Levels in in Peripheral Blood Mononuclear Cells (PBMCs)
Description: During the first cycle (either Cycle 1 non-DDI or Cycle 1-DDI) blood samples will be collected for pharmacodynamic marker assessments by flow cytometry such as phospho-ERK and phospho- S6 activities in PBMCs
Time Frame: DDI cohorts: Days 1, 9 and 10 of Cycle 1; Non-DDI cohorts: Days 1, 8 and 9 of Cycle 1
Population: As the trial was terminated early due to toxicities observed with the combination of pimasertib and temsirolimus, it was decided as per plan not to evaluate the biomarker data for this study
Arm/Group | Pimasertib 45 mg+Temsirolimus 12.5 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (DDI) | Pimasertib 45 mg+Temsirolimus 25 mg (Non-DDI) | Pimasertib 75 mg+Temsirolimus 25 mg (Non-DDI)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the start of the trial treatment until data cut-off date (23 February 2012)
Arm/Group | Pimasertib 45 mg+Temsirolimus 12.5 mg | Pimasertib 45 mg+Temsirolimus 25 mg | Pimasertib 75 mg+Temsirolimus 25 mg
Serious Adverse Events (participants affected / at risk) | 3/4 | 17/23 | 5/6
Other Adverse Events (participants affected / at risk) | 4/4 | 23/23 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pimasertib 45 mg+Temsirolimus 12.5 mg (N=4) | Pimasertib 45 mg+Temsirolimus 25 mg (N=23) | Pimasertib 75 mg+Temsirolimus 25 mg (N=6)
Visual impairment (Eye disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 3 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 3 | 1
Pneumonia (Infections and infestations) | 0 | 4 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Clostridial infection (Infections and infestations) | 0 | 0 | 1
Clostridium difficile sepsis (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Extremity necrosis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pimasertib 45 mg+Temsirolimus 12.5 mg (N=4) | Pimasertib 45 mg+Temsirolimus 25 mg (N=23) | Pimasertib 75 mg+Temsirolimus 25 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 3 | 9 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 4 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 13 | 5
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Chorioretinopathy (Eye disorders) | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0
Detachment of retinal pigment epithelium (Eye disorders) | 0 | 2 | 0
Dry eye (Eye disorders) | 0 | 1 | 0
Eye disorder (Eye disorders) | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 1 | 0
Retinal disorder (Eye disorders) | 0 | 1 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 2 | 0
Visual impairment (Eye disorders) | 0 | 2 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 9 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 3 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 15 | 5
Vomiting (Gastrointestinal disorders) | 0 | 3 | 1
Application site reaction (General disorders) | 0 | 0 | 1
Asthenia (General disorders) | 1 | 2 | 1
Chest discomfort (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 2 | 0
Chills (General disorders) | 1 | 5 | 0
Early satiety (General disorders) | 0 | 2 | 0
Face oedema (General disorders) | 0 | 2 | 0
Fatigue (General disorders) | 2 | 13 | 2
Malaise (General disorders) | 1 | 2 | 1
Oedema peripheral (General disorders) | 1 | 7 | 1
Pyrexia (General disorders) | 2 | 5 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0
Breast infection (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1
Eye infection (Infections and infestations) | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Infusion site infection (Infections and infestations) | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0
lung infection (Infections and infestations) | 0 | 1 | 0
oral candidiasis (Infections and infestations) | 1 | 6 | 0
Paronychia (Infections and infestations) | 0 | 2 | 0
Pharyngitis (Infections and infestations) | 0 | 2 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 4 | 2
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 4 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 6 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 1 | 0
Blood creatinine phosphokinase increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 2 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 1 | 1 | 1
Grip strength decreased (Investigations) | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 9 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 6 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 8 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 2 | 0
Hemianopia homonymous (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0
Myoclonus (Nervous system disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 2 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0
Mental status changes (Psychiatric disorders) | 0 | 2 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 2
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 2 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal fistula (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 8 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 6 | 5
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 4 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
No formal efficacy evaluation was performed for this trial due to early termination of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No